CLINICAL TRIAL: NCT06987604
Title: Continuous Renal Replacement Therapy Intensity in TreatIng Critical Ammonemia Levels
Brief Title: Continuous Renal Replacement Therapy Intensity in Hyperammonemia
Acronym: CRITICAL
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: FIPE - Fundo de Incentivo a Pesquisa do Hospital de Clínicas de Porto Alegre (Unknown)
Responsible Party: Principal Investigator, Gabriel Sartori Pacini, MD, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 88020325.3.1001.5327
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-05

CONDITIONS: Acute Liver Failure; Acute on Chronic Liver Failure (ACLF); Acute Kidney Injury; Ammonia Metabolism
Keywords: ammonia; continuous renal replacement therapy; acute liver failure; acute on chronic liver failure; acute kidney injury
MeSH Terms: conditions — Liver Failure, Acute; Acute-On-Chronic Liver Failure; Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to receive either conventional-dose (25-35 mL/kg/h) or high-dose (45-55 mL/kg/h) continuous renal replacement therapy. Each participant will remain in their assigned treatment arm throughout the study period.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the treatment allocation. Clinical staff and investigators responsible for administering the intervention will not be blinded due to the nature of the dialysis prescription. However, standardized data collection protocols and blinded outcome adjudication will be employed to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Dose CRRT (Experimental): Participants in this group will receive continuous renal replacement therapy (CRRT) at a high effluent dose of 45-55 mL/kg/h for the treatment of hyperammonemia in the context of acute liver failure (ALF) or acute-on-chronic liver failure (ACLF).
  Interventions: Device: High-dose continuous renal replacement therapy
- Conventional-Dose CRRT (Active Comparator): Participants in this group will receive continuous renal replacement therapy (CRRT) at a conventional effluent dose of 25-35 mL/kg/h for the treatment of hyperammonemia in the context of acute liver failure (ALF) or acute-on-chronic liver failure (ACLF).
  Interventions: Device: Conventional-dose continuous renal replacement therapy

INTERVENTIONS:
Device: High-dose continuous renal replacement therapy — Continuous renal replacement therapy administered at an effluent dose of 45-55 mL/kg/h using standard equipment and protocols for critically ill patients with ALF or ACLF and hyperammonemia.
  Arms: High-Dose CRRT
Device: Conventional-dose continuous renal replacement therapy — Continuous renal replacement therapy administered at an effluent dose of 25-35 mL/kg/h using standard equipment and protocols for critically ill patients with ALF or ACLF and hyperammonemia.
  Arms: Conventional-Dose CRRT

SUMMARY:
Acute liver failure (ALF) and acute-on-chronic liver failure (ACLF) are life-threatening conditions often associated with hyperammonemia, hepatic encephalopathy, and multi-organ dysfunction. Ammonia plays a central role in the pathogenesis of cerebral edema and neurotoxicity. Continuous renal replacement therapy (CRRT) has been shown to effectively reduce serum ammonia levels and may improve transplant-free survival in ALF. However, the optimal dialysis dose for ammonia clearance and neurological recovery remains uncertain. This randomized, multicenter clinical trial aims to compare conventional-dose (25-35 mL/kg/h) versus high-dose (45-55 mL/kg/h) CRRT in patients with ALF or ACLF and arterial ammonia >72 μmol/L. The primary outcome is the number of coma- and delirium-free days. Secondary outcomes include ammonia clearance and additional parameters of cerebral function monitoring.

DETAILED DESCRIPTION:
Acute liver failure (ALF) and acute-on-chronic liver failure (ACLF) are critical conditions characterized by rapid deterioration in hepatic function, coagulopathy, hepatic encephalopathy, and multi-organ failure. Elevated serum ammonia levels are frequently observed in these patients and are strongly associated with cerebral dysfunction, including coma and delirium. Ammonia contributes to the development of brain edema through mechanisms involving astrocyte swelling, oxidative stress, and altered neurotransmission. Rapid and effective reduction of ammonia is a key therapeutic target in the management of these patients.

Continuous renal replacement therapy (CRRT) is commonly used in critically ill patients with ALF or ACLF, particularly in those with hyperammonemia. While CRRT is effective in lowering ammonia levels, there is currently no consensus regarding the optimal dialysis dose to maximize ammonia clearance and improve neurological outcomes. Observational data and small interventional studies suggest a potential benefit of higher CRRT doses in terms of ammonia removal and clinical improvement, but robust evidence from randomized trials is lacking.

This study is a randomized, controlled, multicenter clinical trial designed to compare the effects of two different CRRT dosing strategies on cerebral function in patients with ALF or ACLF and arterial ammonia levels >72 μmol/L. Eligible patients will be randomized to receive either conventional-dose CRRT (25-35 mL/kg/h) or high-dose CRRT (45-55 mL/kg/h). All other aspects of clinical management will follow current standard-of-care protocols.

The primary endpoint is the number of coma- and delirium-free days during the intervention period. Secondary outcomes include the degree of ammonia clearance, time to normalization of ammonia levels, filter lifespan, need for rescue therapies (e.g., liver transplantation), mortality, and neurological function monitoring using noninvasive technologies. The study seeks to generate high-quality evidence to guide CRRT dosing decisions in the context of hyperammonemia due to liver failure.

Protocol Amendment - Change in Stratification Ratio The original protocol assumed a balanced enrollment of patients with Acute Liver Failure (ALF) and Acute-on-Chronic Liver Failure (ACLF), with an intended 1:1 distribution across both strata. However, after initiating recruitment and observing actual prevalence patterns at participating centers, it became evident that the number of eligible patients with ACLF significantly exceeds that of ALF.

In response, the study protocol was amended to reflect a revised stratification ratio of 1:5 (ALF: ACLF). Within each stratum, randomization to treatment arms (conventional-dose vs. high-dose CRRT) remains 1:1.

This adjustment enhances recruitment feasibility and reflects the real-world distribution of liver failure phenotypes, without altering the study's scientific objectives, eligibility criteria, or outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of acute liver failure (ALF) or acute-on-chronic liver failure (ACLF) Presence of hyperammonemia, defined as: Arterial ammonia >72 μmol/L and hepatic encephalopathy grade ≥2 or Arterial ammonia >100 μmol/L regardless of encephalopathy grade
* Indication for continuous renal replacement therapy (CRRT), as determined by the attending medical team
* Informed consent provided by the patient or legal representative

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Diagnosis of acute liver failure (ALF) in the context of severe hemodynamic instability
* ALF secondary to ischemic hepatic injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2029-05-14 (Estimated); Study Completion 2029-05-14 (Estimated)

PRIMARY OUTCOMES:
Number of coma- and delirium-free days | Day 1 to Day 28 post-randomization
  The number of days during the first 28 days after randomization in which the patient is alive and free of coma or delirium, assessed using standardized neurological evaluation tools such as the Richmond Agitation-Sedation Scale (RASS) and Confusion Assessment Method for the ICU (CAM-ICU).

SECONDARY OUTCOMES:
Ammonia clearance at 12, 24, 48, and 72 hours | Baseline to 72 hours
  Serial arterial ammonia levels will be measured to calculate the reduction in ammonia concentration from baseline at 12, 24, 48, and 72 hours after initiation of CRRT.
Length of hospital stay | Up to 90 days
  Total number of days from hospital admission to discharge
28-day mortality | 28 days post randomization
  All-cause mortality within 28 days after randomization
90-day mortality | 90 days post-randomization
  All-cause mortality within 90 days after randomization.
Number of ventilator-free days within 28 days | 28 days post-randomization
  Number of days within the first 28 days post-randomization during which the patient is alive and not receiving invasive mechanical ventilation.
Incidence of safety outcomes, such as hypophosphatemia, dialysis disequilibrium syndrome, and rapid correction of hyponatremia | From CRRT initiation up to 7 days or until therapy discontinuation
  Adverse events will be monitored and recorded during CRRT, including laboratory-confirmed hypophosphatemia (phosphate <2.5 mg/dL), clinical signs of dialysis disequilibrium syndrome, and serum sodium correction >10 mmol/L in 24 hours.
Improvement in cerebral compliance | Baseline to Day 28 post-randomization
  Cerebral compliance will be assessed using the Brain4care noninvasive monitoring system. Improvement will be defined as normalization or favorable trend in intracranial compliance waveform patterns compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes